CLINICAL TRIAL: NCT01529905
Title: Longitudinal Study of Individuals Presenting With a First Treated Episode of Depression of Mania (First Episode Project)
Brief Title: Longitudinal Study of People Presenting for First Treatment of a Mood Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Ontario Mental Health Foundation (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 99-1715
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2005-06

CONDITIONS: Major Depression; Bipolar Disorder
Keywords: depression; mania; bipolar; outcome; cognitive
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression; Mania

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The goal of this project is to study the course and outcome of illness in individuals who present with a first episode of depression or mania, or who have a recurrent disorder but have never received treatment. We plan to examine psychological, physical, social and environmental factors that may affect long-term outcome in these disorders

DETAILED DESCRIPTION:
The proposed study is a prospective naturalistic study of patients with a first treated episode of mania or depression. Patients male or female between the ages of 16 and 50 inclusive with a Mood Disorder according to DSM-IV criteria. Control subjects will also be recruited for this study and undergo the same initial testing. Follow-up visits every second year will be requested of control participants.

Patients will be recruited through Family Physicians, and referrals to the Mood Disorders Program. We will respond to referrals with a brief telephone screening interview, and appropriate referrals will be prior to the initiation of medication. Study patients will be treated according to clinic practice guidelines for major depressive disorder and bipolar disorder, as well as for comorbid psychiatric conditions. At intake, a variety of measures will be used to collect data on symptoms and co-morbidity, cognitive processing, social functioning, family and personal history, life events, substance use, mood symptoms, personality functioning and characteristics, and physical well-being (baseline blood work and urine, heart rate, blood pressure, weight).

This study will address issues regarding both structural and functional brain changes that occur in mood disorders by including both imaging and cognitive tests on subjects at entry into the protocol, as well as re-testing with cognitive tests annually and study end-point. Magnetic resonance imaging will be used to obtain data on anatomic structures in the brain. MRI's will be repeated every two years. A small number of subjects (15) from each group of depressed patients (first episode, never treated and multiple past episode patients, never treated) as well as in healthy control subjects will along with the MRI be asked to complete a magnetic resonance spectroscopy (MRS) and a functional MRI.

Episodes of mood elevation and depression will be monitored and recorded with respect to time of onset, level of symptoms, time to remission and recovery, and time to relapse or recurrence if applicable. Subjects will be monitored by clinicians on a regular basis as indicated by their degree of illness and their individual treatment.

In addition to clinical care, all subjects will complete a diagnostic work up which will take approximately 4 hours and include diagnostic, functional, cognitive and physical assessments including routine blood and urine tests. Then weekly visits/contacts for up to one (1) hour in duration for at least eight (8) weeks, then monthly follow-up visits of up to one (1) hour. Brief clinical assessments and self-report questionnaires will be completed at these visits and further blood tests every six months will be required along with weight, waist/hip circumference, blood pressure and pulse rate. Additional blood tests may be required as clinically indicated.

The exact number of visits will depend on the degree of illness and the speed of recovery. Euthymia Testing will be completed after achieving two (2) weeks of Ham-17 ratings less then 7, which will include the following assessments: CVLT, CFQ, MOS, Sub-syndromal Scale, COPE, SAS-R, NEO-PI-R and the "Mood Induction". Annual (on subjects' entry into the study) Testing will be completed; at which time a repeat of the initial assessments will be done. The duration of this study is two years with a possible extension of two more years if the subjects has completed the study requirements and are interested in continuing their participation. Each subject will be asked to complete the final visit(s), which would include a repeat of the initial assessments and a MRI.

Patients who require ongoing clinical care will continue to be followed by their treating psychiatrist following completion of the study protocol. This process will provide a database through which patient characteristics at the time of initial presentation may be examined in relation to the onset and course of illness, prognosis, and response to various forms of treatment. While some of these factors have been examined in previous studies, little information is available on patients who are treatment naive at time of study entry. This project seeks to explore these issues and to provide a basis for further research in the area of first episode mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Primary Mood Disorder,
* Age 16-50
* No previous treatment with psychotropic medication (may have had a max. of 5 days treatment with antidepressants/mood stabilizer &/or they may have Haldol &/or Lorazepam for clear restraint)

Exclusion Criteria:

* History of CNS illness (except migraines),
* Thyroid Disease,
* Neoplastic illness
* History of, or currently being treated for, Anorexia or Bulimia
* History of Traumatic Brain Injury
* Current treatment of Attention-Deficit Hyperactivity Disorder (ADHD)
* Previous diagnosis of OCD or primary Anxiety disorder
* Axis-II diagnosis that would suggest non-responsiveness to pharmacotherapy.
* Substance dependence

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients who present to a tertiary care clinic for first treatment of depression or mania
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 1999-06; Primary Completion 2009-09 (Actual); Study Completion 2014-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Glenda MacQueen, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, Centre for Mountain Health Services, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Judd LL, Akiskal HS, Maser JD, Zeller PJ, Endicott J, Coryell W, Paulus MP, Kunovac JL, Leon AC, Mueller TI, Rice JA, Keller MB. A prospective 12-year study of subsyndromal and syndromal depressive symptoms in unipolar major depressive disorders. Arch Gen Psychiatry. 1998 Aug;55(8):694-700. doi: 10.1001/archpsyc.55.8.694. PMID 9707379
- [Background] Solomon DA, Keller MB, Leon AC, Mueller TI, Shea MT, Warshaw M, Maser JD, Coryell W, Endicott J. Recovery from major depression. A 10-year prospective follow-up across multiple episodes. Arch Gen Psychiatry. 1997 Nov;54(11):1001-6. doi: 10.1001/archpsyc.1997.01830230033005. PMID 9366656
- [Background] Mueller TI, Keller MB, Leon AC, Solomon DA, Shea MT, Coryell W, Endicott J. Recovery after 5 years of unremitting major depressive disorder. Arch Gen Psychiatry. 1996 Sep;53(9):794-9. doi: 10.1001/archpsyc.1996.01830090040006. PMID 8792756